CLINICAL TRIAL: NCT02083575
Title: Study of Safty and Efficacy of Adjuvant Vitamin c in Augmenting Iron Chelation
Brief Title: Role of Vitamin C to Augment Iron Chelation With DFP or DFX
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: vitamin c and iron chelator
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Vitamin c; Thalassemia Major; Iron Chelation
Keywords: vitamin c; thalassemia major; iron chelation
MeSH Terms: conditions — beta-Thalassemia | interventions — Ascorbic Acid; Isoflurophate; Deferiprone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin c (Active Comparator): 25 heavily iron-loaded thalassemia patients, receiving adjuvant vitamin c with iron chelator.
  Interventions: Drug: Vitamin C, Defriprone, deferisarox
- iron chelator (Other): Included 25 heavily iron-loaded thalassemia patients, not receiving adjuvant vitamin c with iron chelator.
  Interventions: Drug: deferiprone , deferesarox

INTERVENTIONS:
Drug: Vitamin C, Defriprone, deferisarox — adjuvant vitamin c with iron chelator.
  Other Names: vitamin c; DFP; DFX
  Arms: vitamin c
Drug: deferiprone , deferesarox — iron chelator
  Other Names: DFP; DFX
  Arms: iron chelator

SUMMARY:
role of Vit C to Augment iron chelation with DFP or DFX in thalassemic patients.

DETAILED DESCRIPTION:
assess safety and efficacy of Vit C to Augment iron chelation with DFP or DFX in thalassemic patients.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with overload secondary to thalassemia major

Exclusion Criteria:

* • with HIV positive or have active HCV.

  * A history of serious immunologic hypersensitivity to any medication such as anaphylaxis or angioedema.
  * Participation in a previous investigational drug study within the 30 days preceding screening.
  * A woman of childbearing potential must have a negative serum pregnancy test at screening. She must use a medically acceptable form of birth control during the study and for a month afterwards who are pregnant or breast-feeding.
  * An inability to adhere to the designated procedures and restrictions of this protocol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Vit C to Augment iron chelation | 12 months
  assess safety and efficacy of Vit C to Augment iron chelation with DFP or DFX in thalassemic patients.
vitamin c augmenting effect of iron chelator | 12 month
  better reduction in serum ferritin, LIC and cardiac T28 in group receiving vitamin c

SECONDARY OUTCOMES:
adverse related events | 12 month
  safety and occurrence of AEs in both studied groups

CONTACTS AND LOCATIONS:
Overall Officials: MOHSEN S ELALFY, PROF., Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Hematology clinic, Ain Shams University Egypt, Cairo, Egypt